CLINICAL TRIAL: NCT00078403
Title: Suppressive Long-Term Antiviral Management of Hepatitis C Virus (HCV) and HIV-1 Coinfected Subjects (SLAM-C)
Brief Title: Pegylated Interferon Alfa-2a Maintenance Therapy and Liver Disease Progression in People Infected With Both HIV and Hepatitis C Virus (HCV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5178; 10008 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2004-02-24; First posted 2004-02-25 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2016-11

CONDITIONS: HIV Infections; Hepatitis C; Liver Disease
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hepatitis C; Liver Diseases | interventions — peginterferon alfa-2a; Ribavirin

ARMS (3):
- Arm A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) (Experimental): At week 12 (end of the initial run-in period - Step 1) participants were found to have detectable HCV RNA (HCV RNA >=600 IU/mL) and had less than a 2 log10 decrease in HCV RNA from baseline. For Step 2, participants were randomized to receive the pegylated interferon (PEG-IFN) 180 mcg weekly for 72 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Arm B: OL (PEG-IFN, RBV) then OL Randomized (Observation) (Experimental): At week 12 (end of the initial run-in period - Step 1) participants were found to have detectable HCV RNA (HCV RNA >=600 IU/mL) and had less than a 2 log10 decrease in HCV RNA from baseline. For Step 2, participants were randomized to 72 weeks of observation (no treatment).
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Arm C: OL (PEG-IFN, RBV) then OL (PEG-IFN, RBV) (Experimental): At week 12 (end of initial run-in period, Step 1) participants were found to have undetectable HCV RNA (HCV RNA <600 IU/mL) or at least a 2 log10 decrease in HCV RNA from baseline. Participants entered Step 3 and were assigned to continue the run-in treatment (PEG-IFN 180 mcg weekly & RBV1-1.2 g/day based on weight) for a total of 72 weeks. At week 36, participants who had detectable HCV RNA (HCV RNA >=60 IU/mL using a qualitative assay) could enter Step 2 and be randomized to OL PEG-IFN or Observation.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 180 mcg PEG-IFN subcutaneously
Drug: Ribavirin — One tablet or capsule containing ribavirin 200 mg

SUMMARY:
Infection with both HIV and hepatitis C virus (HCV) may result in serious and sometimes fatal liver disease. The purpose of this study was to test the effectiveness of long-term pegylated interferon alfa-2a (PEG-IFN) and ribavirin treatment in slowing liver disease progression in people infected with both HIV and HCV.

DETAILED DESCRIPTION:
Rapid progression of liver disease to liver failure has been observed in people coinfected with HIV and HCV. This observation appears to be directly related to an increase in the rate of fibrotic progression in the liver compared to people infected with HCV alone. PEG-IFN and ribavirin are used in standard treatment of HCV. This study tested the effectiveness of using PEG-IFN in reducing the rate of liver fibrosis progression in participants coinfected with HIV and HCV who could not lower their HCV viral load to undetectable or who could not maintain their HCV viral load at undetectable on PEG-IFN and ribavirin treatment.

Participants entered Step 1 (initial run-in period) to receive 12 weeks of 180 mcg PEG-IFN subcutaneously once weekly plus 1 to 1.2 g/day ribavirin based on body weight. At week 12, HCV RNA testing was performed.

Participants with early virologic response (EVR), defined as >=2 log10 drop in HCV RNA from baseline or undetectable HCV RNA (<600 IU/ml with quantitative assay used in Step 1) at Week 12, who had tolerated Step 1 treatment, entered into Step 3 to continue receiving the Step 1 treatment for a total of 72 weeks (Arm C). Participants who did not meet the criteria for entry into Step 3 were discontinued from the study. In Step 3, participants were followed for an additional 24 weeks after treatment discontinuation to determine sustained virologic response (SVR). Initially, Step 3 participants who had a detectable HCV viral load (>=60 IU/ml with the qualitative assay used in Step 3) at Week 36 were eligible to enroll in Step 2. After early closure of Step 2, such participants remained in Step 3 until study completion.

Participants with <2 log10 drop in HCV RNA from baseline and detectable HCV RNA at Week 12 (non-EVR) discontinued Step 1 treatment. Non-EVRs who met the Step 2 eligibility criteria, were enrolled in Step 2 and randomized to receive 180 mcg PEG-IFN subcutaneously weekly for 72 weeks (Arm A) or observation for 72 weeks (Arm B). Participants who did not meet the criteria for entry into Step 2 were discontinued from the study. Step 2 of the study was closed prematurely in May 2007 due to lower than expected progression rates among the participants in the observation arm such that the primary objective could not be reached. There were no safety concerns.

Liver biopsies were conducted at study screening, and at Step 2 entry and exit until the early closure of Step 2. Medical history assessment, physical exams, and blood collection were conducted every 4-12 weeks for participants in Steps 1, 2, and 3. Participants were followed for up to 18 weeks in Step 1, followed by a total of 72 in Step 2 or by up to a total of 84 weeks in Step 3.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* HIV infected
* Stable antiretroviral therapy for at least 8 weeks prior to study entry OR have not received any antiretroviral therapy for at least 4 weeks prior to entry
* HIV viral load less than 50,000 copies/ml within 6 weeks prior to study entry
* CD4 count greater than 200 cells/mm^3 within 6 weeks prior to study entry
* Hepatitis C virus (HCV) infected
* Either HCV treatment naive OR previously treated with interferon (IFN), PEG-IFN, IFN and ribavirin, or PEG-IFN and ribavirin for at least 12 weeks and HCV RNA positive following their last course of HCV treatment
* Chronic liver disease consistent with chronic viral hepatitis
* At least stage I fibrosis on a liver biopsy obtained within 104 weeks of study entry
* If at stage VI fibrosis, Child-Pugh-Turcotte (CPT) score of 5 or less and no more than Child-Pugh Class A
* Liver enzyme (alanine aminotransferase [ALT], aspartate aminotransferase [AST], and alkaline phosphatase) levels 10 times or less than upper limit of normal
* Agree to use acceptable methods of contraception

Inclusion Criteria for Step 2:

* Currently enrolled in Step 1 or received 12 weeks of PEG-IFN plus ribavirin outside this study
* Detectable HCV viral load and <2 log10 decrease from baseline in plasma/serum HCV viral load at Week 12.
* On Step 1 study treatment for no longer than 18 weeks

Inclusion Criteria for Step 3:

* Currently enrolled in Step 1
* Undetectable HCV RNA or a 2-log or greater decrease in plasma/serum HCV viral load.
* On Step 1 study treatment for no longer than 18 weeks

Exclusion Criteria for Steps 1 and 3:

* Have received HCV treatment within 4 weeks of study entry. Participants currently receiving treatment for HCV, if non-EVRs, were considered for direct entry into Step 2, without the run-in period in Step 1.
* Could not tolerate treatment with PEG-IFN, defined as missing 3 or more consecutive PEG-IFN doses during the first 12 weeks or a total of 5 doses prior to Step 3 entry. Participants who have missed doses of ribavirin will not be excluded from Step 3 entry.
* Use of granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 14 days prior to study entry
* Alpha feto protein level 400 ng/ml or greater within 24 weeks prior to study entry, or alpha feto protein level greater than 50 ng/ml and less than 400 ng/ml (unless computed tomography [CT] scan or magnetic resonance imaging [MRI] shows no evidence of hepatic tumor) within 24 weeks prior to study entry
* Decompensated liver disease, including presence or history of ascites, variceal bleeding, and brain or nervous system damage as a result of liver damage
* Other causes of significant liver disease, including hepatitis A or B, excess iron deposits in the liver (hemochromatosis), or homozygote alpha-1 antitrypsin deficiency
* Use of systemic corticosteroids, interferon gamma, TNF-alpha inhibitors, rifampin, rifabutin, pyrazinamide, isoniazid, ganciclovir, or hydroxyurea within 2 weeks prior to study entry
* Known allergy/sensitivity to PEG-IFN alfa-2a or ribavirin or their formulations
* History of uncontrolled seizure disorders
* Clinically active thyroid disease. Thyroid hormone replacement therapy is permitted, but thyroid-stimulating hormone (TSH) and free thyroxine index (FTI) must be in normal range.
* History of autoimmune processes, including Crohn's disease, ulcerative colitis, severe psoriasis, and rheumatoid arthritis, that may be made worse by interferon use
* Any systemic antineoplastic or immunomodulatory treatment or radiation within 24 weeks prior to study entry
* Malignancy
* Active coronary artery disease within 24 weeks prior to study entry
* Acute or active AIDS-defining opportunistic infections within 12 weeks of study entry
* Hemoglobin abnormalities (e.g., thalassemia) or any other cause of or tendency to break down red blood cells (hemolysis)
* History of major organ transplantation with an existing functional graft
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with study adherence
* Uncontrolled or active depression or other psychiatric disorder, such as untreated Grade 3 psychiatric disorder, medically untreatable Grade 3 disorder, or any hospitalization within 52 weeks of study entry that, in the opinion of the investigator, may interfere with study requirements
* Other serious illness or chronic medical condition that, in the opinion of the investigator, may have prevented participant's completion of the study
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2004-07; Primary Completion 2007-05 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E. Sherman, MD, PhD, Study Chair — University of Cincinnati; Raymond Chung, MD, Study Chair — Harvard/Massachusetts General Hospital
Locations (37):
- United States (36):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - University of Southern California CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Weill Cornell Chelsea CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Trillium Health ACTG CRS, Rochester, New York
  - McCree McCuller Wellness Ctr. at the Connection, Infectious Disease Unit, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Cincinnati CRS, Cincinnati, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Univ. of Pennsylvania Health System, Presbyterian Med. Ctr., Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Univ. of Texas Southwestern Med. Ctr., Amelia Court Continuity Clinic, Dallas, Texas
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Brau N. Treatment of chronic hepatitis C in human immunodeficiency virus/hepatitis C virus-coinfected patients in the era of pegylated interferon and ribavirin. Semin Liver Dis. 2005 Feb;25(1):33-51. doi: 10.1055/s-2005-864780. PMID 15731996
- [Background] Borgia G, Reynaud L, Gentile I, Piazza M. HIV and hepatitis C virus: facts and controversies. Infection. 2003 Aug;31(4):232-40. doi: 10.1007/s15010-003-3131-4. PMID 14562947
- [Background] Khalili M, Bernstein D, Lentz E, Barylski C, Hoffman-Terry M. Pegylated interferon alpha-2a with or without ribavirin in HCV/HIV coinfection: partially blinded, randomized multicenter trial. Dig Dis Sci. 2005 Jun;50(6):1148-55. doi: 10.1007/s10620-005-2723-5. PMID 15986873
- [Background] Neau D, Trimoulet P, Winnock M, Rullier A, Le Bail B, Lacoste D, Ragnaud JM, Bioulac-Sage P, Lafon ME, Chene G, Dupon M; ROCO Study Group. Comparison of 2 regimens that include interferon-alpha-2a plus ribavirin for treatment of chronic hepatitis C in human immunodeficiency virus-coinfected patients. Clin Infect Dis. 2003 Jun 15;36(12):1564-71. doi: 10.1086/375067. Epub 2003 Jun 3. PMID 12802757
- [Background] Torriani FJ, Ribeiro RM, Gilbert TL, Schrenk UM, Clauson M, Pacheco DM, Perelson AS. Hepatitis C virus (HCV) and human immunodeficiency virus (HIV) dynamics during HCV treatment in HCV/HIV coinfection. J Infect Dis. 2003 Nov 15;188(10):1498-507. doi: 10.1086/379255. Epub 2003 Nov 13. PMID 14624375
- [Background] Torriani FJ, Rodriguez-Torres M, Rockstroh JK, Lissen E, Gonzalez-Garcia J, Lazzarin A, Carosi G, Sasadeusz J, Katlama C, Montaner J, Sette H Jr, Passe S, De Pamphilis J, Duff F, Schrenk UM, Dieterich DT; APRICOT Study Group. Peginterferon Alfa-2a plus ribavirin for chronic hepatitis C virus infection in HIV-infected patients. N Engl J Med. 2004 Jul 29;351(5):438-50. doi: 10.1056/NEJMoa040842. PMID 15282351
- [Background] The Division of AIDS Table for Grading the Severity of Adult Adverse Events (DAIDS AE Grading Table), August 1992.
- [Background] Manual for Expedited Reporting of Adverse Events to Division of AIDS (DAIDS EAE Manual), May 2004.
- [Result] Butt AA, Umbleja T, Andersen JW, Chung RT, Sherman KE; ACTG A5178 Study Team. The incidence, predictors and management of anaemia and its association with virological response in HCV / HIV coinfected persons treated with long-term pegylated interferon alfa 2a and ribavirin. Aliment Pharmacol Ther. 2011 Jun;33(11):1234-44. doi: 10.1111/j.1365-2036.2011.04648.x. Epub 2011 Mar 29. PMID 21535051
- [Result] Sherman KE, Andersen JW, Butt AA, Umbleja T, Alston B, Koziel MJ, Peters MG, Sulkowski M, Goodman ZD, Chung RT; AIDS Clinical Trials Group A5178 Study Team. Sustained long-term antiviral maintenance therapy in HCV/HIV-coinfected patients (SLAM-C). J Acquir Immune Defic Syndr. 2010 Dec 15;55(5):597-605. doi: 10.1097/QAI.0b013e3181f6d916. PMID 20921898
- [Result] Chung RT, Umbleja T, Chen JY, Andersen JW, Butt AA, Sherman KE; Actg A5178 Study Team. Extended therapy with pegylated interferon and weight-based ribavirin for HCV-HIV coinfected patients. HIV Clin Trials. 2012 Mar-Apr;13(2):70-82. doi: 10.1310/hct1302-70. PMID 22510354
- [Result] Butt AA, Umbleja T, Andersen JW, Sherman KE, Chung RT; ACTG A5178 Study Team. Impact of peginterferon alpha and ribavirin treatment on lipid profiles and insulin resistance in Hepatitis C virus/HIV-coinfected persons: the AIDS Clinical Trials Group A5178 Study. Clin Infect Dis. 2012 Sep;55(5):631-8. doi: 10.1093/cid/cis463. Epub 2012 May 4. PMID 22563020
- [Derived] Branch AD, Kang M, Hollabaugh K, Wyatt CM, Chung RT, Glesby MJ. In HIV/hepatitis C virus co-infected patients, higher 25-hydroxyvitamin D concentrations were not related to hepatitis C virus treatment responses but were associated with ritonavir use. Am J Clin Nutr. 2013 Aug;98(2):423-9. doi: 10.3945/ajcn.112.048785. Epub 2013 Jun 5. PMID 23739141
- [Derived] Shire NJ, Rao MB, Succop P, Buncher CR, Andersen JA, Butt AA, Chung RT, Sherman KE; AIDS Clinical Trials Group 5178 Study Group. Improving noninvasive methods of assessing liver fibrosis in patients with hepatitis C virus/human immunodeficiency virus co-infection. Clin Gastroenterol Hepatol. 2009 Apr;7(4):471-80, 480.e1-2. doi: 10.1016/j.cgh.2008.12.016. Epub 2008 Dec 25. PMID 19268724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: People with hepatitis C virus (HCV)/HIV coinfection were recruited for participation in this study.
Pre-assignment Details: 330 participants were to receive 12 weeks of PEG+RBV to determine EVR status. Of the 330, 33 discontinued prior to week 12; 113 were non-EVRs, 80 of whom were randomized between Arms A and B; and 184 achieved EVR, 170 of whom were eligible to continue. 169 of the 170 were assigned to Arm C and one was inadvertently randomized between Arms A and B.
Groups:
- Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN): At week 12 (end of the initial run-in period - Step 1) participants were found to have detectable HCV RNA (HCV RNA >=600 IU/mL) and had less than a 2 log10 decrease in HCV RNA from baseline. For Step 2, participants were randomized to receive the pegylated interferon (PEG-IFN) 180 mcg weekly for 72 weeks.
- OL (PEG-IFN, RBV) Then OL Randomized (Observation): At week 12 (end of the initial run-in period - Step 1) participants were found to have detectable HCV RNA (HCV RNA >=600 IU/mL) and had less than a 2 log10 decrease in HCV RNA from baseline. For Step 2, participants were randomized to 72 weeks of observation (no treatment).
- OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV): At week 12 (end of initial run-in period, Step 1) participants were found to have undetectable HCV RNA (HCV RNA <600 IU/mL) or at least a 2 log10 decrease in HCV RNA from baseline. Participants entered Step 3 and were assigned to continue the run-in treatment (PEG-IFN 180 mcg weekly & RBV1-1.2 g/day based on weight) for a total of 72 weeks. At week 36, participants who had detectable HCV RNA (HCV RNA >=60 IU/mL using a qualitative assay) could enter Step 2 and be randomized to OL PEG-IFN or Observation.
Period: Overall Study
Arm/Group | Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | OL (PEG-IFN, RBV) Then OL Randomized (Observation) | OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Started | 44 (Eligible at pre-assignment (40), direct (2), Arm C week 36 non-response (1), EVR inadvertently (1).) | 42 (Eligible at pre-assignment (40), direct (1), Arm C week 36 non-response (1).) | 169
Completed | 26 | 26 | 141
Not Completed | 18 | 16 | 28

BASELINE CHARACTERISTICS:
Population: All Arm A, B and C participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | OL (PEG-IFN, RBV) Then OL Randomized (Observation) | OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV) | Total
Number analyzed (Participants) | 44 | 42 | 169 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 42 | 169 | 255
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (6.7) | 48.1 (5.8) | 47.2 (7.1) | 47.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 19 | 43
  Male | 32 | 30 | 150 | 212
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 168 | 249
  Puerto Rico | 3 | 2 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time-scaled Change in Metavir Liver Fibrosis Score (SCMFS)
Description: SCMFS is the difference between the Metavir fibrosis scores of the study exit and study entry liver biopsies where the difference is scaled to one year. The SCMFS assesses the annualized change in the severity of liver fibrosis on a continuous scale from -4.0 Metavir units per year (reduced fibrosis over time, a positive study outcome) to +4.0 Metavir units per year (increased fibrosis over time).
Time Frame: Baseline and at week 72 or premature discontinuation
Population: 62 Arm A and B participants who had follow-up liver biopsy performed or those who had Week 72 potential as of May 2, 2007 but no follow-up liver biopsy. In the unadjusted ITT analysis, the participants without SCMFS available were assigned the highest SCMFS (+2).
Measure: Median (Inter-Quartile Range); unit: Metavir units per one year (52 weeks)
Groups:
- A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN): At week 12 (end of the initial run-in period - Step 1) participants were found to have detectable HCV RNA (HCV RNA >=600 IU/mL) and had less than a 2 log10 decrease in HCV RNA from baseline. For Step 2, participants were randomized to receive the pegylated interferon (PEG-IFN) 180 mcg weekly for 72 weeks.
- B: OL (PEG-IFN, RBV) Then OL Randomized (Observation): At week 12 (end of the initial run-in period - Step 1) participants were found to have detectable HCV RNA (HCV RNA >=600 IU/mL) and had less than a 2 log10 decrease in HCV RNA from baseline. For Step 2, participants were randomized to 72 weeks of observation (no treatment).
- C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV): At week 12 (end of initial run-in period, Step 1) participants were found to have undetectable HCV RNA (HCV RNA <600 IU/mL) or at least a 2 log10 decrease in HCV RNA from baseline. Participants entered Step 3 and were assigned to continue the run-in treatment (PEG-IFN 180 mcg weekly & RBV1-1.2 g/day based on weight) for a total of 72 weeks. At week 36, participants who had detectable HCV RNA (HCV RNA >=60 IU/mL using a qualitative assay) could enter Step 2 and be randomized to OL PEG-IFN or Observation.
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 33 | 29 | 0
Metavir units per one year (52 weeks) | 0 [0 to 1.37] | 0 [0 to 2] |
Statistical Analysis 1: Comparison: A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) vs B: OL (PEG-IFN, RBV) Then OL Randomized (Observation); Accrual and follow-up on Arms A and B were halted for futility at the first independent interim review of the primary endpoint conducted on May 2, 2007; Test type: Superiority or Other; p = 0.58, Exact Wilcoxon rank sum test — P-value is pre-specified 1-sided test that PEG slows liver fibrosis progression. Accrual and follow-up on Arms A and B were halted at interim review for lack of fibrosis progression in Arm B (control arm). P-value is unadjusted for interim analysis

2. Secondary Outcome: Number of Participants With Detectable HCV Viral Load (>= 60 IU/mL)
Description: Qualitative plasma HCV viral load was categorized as less than 60 IU/mL vs greater than or equal to 60 IU/mL where 60 IU/mL is the lower limit of qualitative assay used in Steps 2 and 3.
Time Frame: Arms A and B: Weeks 0, 12, 24, 48 and 72; Arm C: Weeks 0, 12, 24, 36, 60, 72, 84
Population: All Arm A, B and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Week 0--Number of participants with HCV RNA data | 44 | 42 | 164
  Week 0--Number of participants with detectable HCV | 42 | 42 | 53
  Week 12--Number of participants with HCV RNA data | 42 | 34 | 158
  Week 12-Number of participants with detectable HCV | 40 | 34 | 31
  Week 24--Number of participants with HCV RNA data | 36 | 35 | 163
  Week 24-Number of participants with detectable HCV | 35 | 35 | 39
  Week 36--Number of participants with HCV RNA data | 0 | 0 | 158
  Week 36-Number of participants with detectable HCV | NA — Test not specified in protocol at this time point. | NA — Test not specified in protocol at this time point. | 41
  Week 48--Number of participants with HCV RNA data | 31 | 28 | 0
  Week 48-Number of participants with detectable HCV | 31 | 28 | NA — Test not specified in protocol at this time point.
  Week 60--Number of participants with HCV RNA data | 0 | 0 | 137
  Week 60-Number of participants with detectable HCV | NA — Test not specified in protocol at this time point. | NA — Test not specified in protocol at this time point. | 34
  Week 72--Number of participants with HCV RNA data | 27 | 22 | 135
  Week 72-Number of participants with detectable HCV | 27 | 22 | 51
  Week 84--Number of participants with HCV RNA data | 0 | 0 | 137
  Week 84-Number of participants with detectable HCV | NA — Test not specified in protocol at this time point. | NA — Test not specified in protocol at this time point. | 50

3. Secondary Outcome: Time-scaled Change in Ishak Liver Inflammation Score (SCIIS)
Description: Liver biopsies were performed within 42 days prior to randomization between Arms A and B while the participant remained on PEG-IFN plus RBV (=entry biopsy) and again at week 72 or premature study discontinuation (=exit biopsy). SCIIS was defined as the difference between the Ishak inflammation score of the exit biopsy and the Ishak inflammation score of the entry biopsy, where the difference is scaled to one year.
Time Frame: Baseline and at week 72 or premature discontinuation
Population: All participants with SCIIS available (Complete Cases)
Measure: Median (Inter-Quartile Range); unit: Ishak units per one year (52 weeks)
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 0
Ishak units per one year (52 weeks) | 0 [-0.75 to 1.79] | 1.31 [0 to 2.10] |

4. Secondary Outcome: Number of Participants With Anemia
Description: Number of participants with anemia by grade (defined by hemoglobin level in grams per deciliter; g/dL). DAIDS Toxicity Grading Table (1992) was used for grading where Grade 1 = hemoglobin of 8 to 9.4 g/dl; Grade 2 = 7 to 7.9 g/dl; Grade 3 = 6.5 to 6.9 g/dl; Grade 4 = below 6.5 g/dl.
Time Frame: Up to 96 weeks
Population: All Arm A, B and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Anemia >= Grade 2 | 1 | 0 | 6
  Grade 2 | 0 | 0 | 3
  Grade 3 | 0 | 0 | 1
  Grade 4 | 1 | 0 | 2

5. Secondary Outcome: Number of Participants With Neutropenia
Description: Number of participants with neutropenia by grade (defined by absolute neutrophil count [ANC] per cubic millimeter; mm^3). DAIDS Toxicity Grading Table (1992) was used for grading where Grade 1 = ANC of 1000 to 1500 /mm^3; Grade 2 = 750 to 999 /mm^3; Grade 3 = 500 to 749 /mm^3; Grade 4 = below 500 /mm^3.
Time Frame: Up to 96 weeks
Population: All Arm A, B and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Neutropenia >= Grade 2 | 20 | 10 | 96
  Grade 2 | 7 | 4 | 38
  Grade 3 | 10 | 5 | 37
  Grade 4 | 3 | 1 | 21

6. Secondary Outcome: Number of Participants With Thrombocytopenia
Description: Number of participants with thrombocytopenia by grade (defined by platelet count per cubic millimeter; mm^3). DAIDS Toxicity Grading Table (1992) was used for grading where Grade 1 = platelets of 75,000 to 99,000 /mm^3; Grade 2 = 50,000 to 74,999 /mm^3; Grade 3 = 20,000 to 49,999 /mm^3; Grade 4 = below 20,000 /mm^3.
Time Frame: Up to 96 weeks
Population: All Arm A, B and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Thrombocytopenia >= Grade 2 | 14 | 4 | 31
  Grade 2 | 10 | 3 | 25
  Grade 3 | 4 | 1 | 5
  Grade 4 | 0 | 0 | 1

7. Secondary Outcome: Number of Participants With Depression and/or Other Psychological Events
Description: Depression and other psychological events. DAIDS Toxicity Grading Table (1992) was used for grading. The protocol required reporting of depression and other psychological events of Grade 3 or higher or if led to a change in treatment, regardless of grade.
Time Frame: Up to 96 weeks
Population: All Arm A, B and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Any psychological | 3 | 1 | 19
  Grade 3 | 2 | 1 | 18
  Grade 4 | 1 | 0 | 1

8. Secondary Outcome: Number of Participants With High-grade Signs and Symptoms or Laboratory Values
Description: Number of participants with high-grade (Grade 3 or higher) signs and symptoms or laboratory values. DAIDS Toxicity Grading Table (1992) was used for grading where Grade 1 = transient/mild discomfort, no limitation in activity, no medical intervention; Grade 2 = mild/moderate limitation in activity, some assistance, no/minimal medical intervention; Grade 3 = marked limitation in activity, some assistance, medical intervention required); Grade 4 = extreme limitation in activity, significant medical intervention, assistance, hospitalization.
Time Frame: Up to 96 Weeks
Population: All Arm A, B and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Any Grade 3 or higher | 22 | 20 | 84
  Grade 3 | 15 | 15 | 73
  Grade 4 | 7 | 5 | 11

9. Secondary Outcome: Number of Participants With Dose Modifications, Temporary Stops, and Premature Treatment Discontinuations
Description: 3-level categorical of the worst of 1) premature treatment discontinuation, 2) temporary stop or 3) dose reduction. For Arm C, the worst for either PEG-IFN or RBV is summarized.
Time Frame: Up to 96 Weeks
Population: All Arm A and C participants. Arm B participants did not receive treatment.
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 0 | 169
Participant
  Premature treatment discontinuation | 16 |  | 57
  Temporarily off treatment | 7 |  | 29
  Reduced dose | 2 |  | 33

10. Secondary Outcome: Number of Participants Adherent to Study Medications
Description: A categorical variable with levels adherent and non-adherent based on participants' self report. For Arm A, adherence was defined as not missing PEG within 2 weeks of visit. For Arm C, adherence was defined as not missing any PEG within 2 weeks of visit and not missing RBV within 4 days of visit.
Time Frame: Arm A: at weeks 12, 24, 48 and 72. Arm C: at entry and weeks 12, 24, 48, 60.
Population: All Arm A and Arm C participants. Arm B participants did not receive treatment.
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 0 | 159
Participant
  Week 0: Number of participants with adherence data | 0 |  | 158
  Week 0: Number of participants adherent to meds | NA — Evaluation not specified in protocol at this timepoint. |  | 132
  Week 12:Number of participants with adherence data | 37 |  | 150
  Week 12:Number of participants adherent to meds | 32 |  | 125
  Week 24:Number of participants with adherence data | 32 |  | 145
  Week 24:Number of participants adherent to meds | 28 |  | 118
  Week 48:Number of participants with adherence data | 22 |  | 120
  Week 48:Number of participants adherent to meds | 19 |  | 95
  Week 60:Number of participants with adherence data | 0 |  | 91
  Week 60:Number of participants adherent to meds | NA — Evaluation not specified in protocol at this timepoint. |  | 79
  Week 72:Number of participants with adherence data | 8 |  | 0
  Week 72:Number of participants adherent to meds | 7 |  | NA — Evaluation not specified in protocol at this timepoint.

11. Secondary Outcome: HCV Polymorphisms
Description: Due to premature closure of Arms A and B with insufficient number of participants for analysis, this outcome measure was not pursued.
Time Frame: Entry and week 72 (Arms A and B only).
Population: Due to premature closure of Arms A and B with insufficient number of participants for analysis, this outcome measure was not pursued. No participants were analyzed.
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: HCV-specific Immune Response in Intrahepatic Lymphocytes
Description: as for outcome 11
Time Frame: Entry and week 72 (Arms A and B only).
Population: as for outcome 11
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With Undetectable HIV Viral Load (<50 Copies/mL)
Description: A blood sample was drawn to determine the HIV-1 viral load. HIV-1 viral load was categorized as <50 copies/mL (undetectable) or >=50 copies/mL (detectable). 50 is the lower limit of detection of the assay.
Time Frame: Arms A and B: Weeks 0, 24, 48 and 72; Arm C: Weeks 0, 12, 24, 36, 48, 60, 72, 84
Population: All Arm A, B, and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Week 0: Number of participants with HIV RNA data | 44 | 42 | 169
  Week 0: No. of participants with undetectable VL | 32 | 34 | 146
  Week 12: Number of participants with HIV RNA data | 0 | 0 | 164
  Week 12: No. of participants with undetectable VL | NA — Test not specified in protocol at this timepoint. | NA — Test not specified in protocol at this timepoint. | 138
  Week 24: Number of participants with HIV RNA data | 39 | 39 | 165
  Week 24: No. of participants with undetectable VL | 25 | 25 | 141
  Week 36: Number of participants with HIV RNA data | 0 | 0 | 160
  Week 36: No. of participants with undetectable VL | NA — Test not specified in protocol at this timepoint. | NA — Test not specified in protocol at this timepoint. | 134
  Week 48: Number of participants with HIV RNA data | 35 | 33 | 150
  Week 48: No. of participants with undetectable VL | 24 | 25 | 125
  Week 60: Number of participants with HIV RNA data | 0 | 0 | 140
  Week 60: No. of participants with undetectable VL | NA — Test not specified in protocol at this timepoint. | NA — Test not specified in protocol at this timepoint. | 113
  Week 72: Number of participants with HIV RNA data | 27 | 27 | 140
  Week 72: No. of participants with undetectable VL | 19 | 20 | 107
  Week 84: Number of participants with HIV RNA data | 0 | 0 | 136
  Week 84: No. of participants with undetectable VL | NA — Test not specified in protocol at this timepoint. | NA — Test not specified in protocol at this timepoint. | 108

14. Secondary Outcome: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: Insulin resistance was evaluated by HOMA-IR, calculated as [fasting glucose (mg/dL) x fasting insulin (uIU/mL)]/405. Study protocol required fasting for at least 8 hours (nothing by mouth except medications and water) prior to specimen collection for fasting insulin and fasting glucose testing.
Time Frame: Arms A and B: at entry and weeks 24, 48 and 72; Arm C: at entry and at weeks 12, 24, 36, 48, 72, 84 and 96.
Population: All Arm A, B and C participants who had HOMA-IR result available. In Arm C, metabolic testing was only performed on participants who enrolled under protocol version 1.0. The number of participants with results available at time points listed in the Time Frame are shown in the Data Table Row Titles below.
Measure: Median (Inter-Quartile Range); unit: mg/dL x uIU/mL
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 98
mg/dL x uIU/mL
  Week 0: HOMA-IR (N=32 in A, 32 in B, 72 in C) | 3.84 [2.77 to 9.03] | 2.49 [1.83 to 4.48] | 2.37 [1.50 to 5.36]
  Week 12: HOMA-IR (N=72 in C) | NA [NA to NA] — HOMA-IR was not collected at Week 12 in Arms A and B. | NA [NA to NA] — HOMA-IR was not collected at Week 12 in Arms A and B. | 2.47 [1.63 to 4.22]
  Week 24: HOMA-IR (N=34 in A, 30 in B, 73 in C) | 3.08 [1.68 to 5.59] | 4.78 [1.78 to 6.13] | 2.58 [1.35 to 4.44]
  Week 36: HOMA-IR (N=66 in C) | NA [NA to NA] — HOMA-IR was not collected at Week 36 in Arms A and B. | NA [NA to NA] — HOMA-IR was not collected at Week 36 in Arms A and B. | 2.41 [1.44 to 4.58]
  Week 48: HOMA-IR (N=30 in A, 24 in B, 74 in C) | 3.53 [1.72 to 6.65] | 2.84 [1.78 to 6.38] | 3.25 [1.73 to 5.01]
  Week 72: HOMA-IR (N=67 in C) | 4.79 [3.41 to 7.83] | 4.82 [2.46 to 9.12] | 2.69 [1.66 to 5.47]
  Week 84: HOMA-IR (N=63 in C) | NA [NA to NA] — HOMA-IR was not collected at Week 84 in Arms A and B. | NA [NA to NA] — HOMA-IR was not collected at Week 84 in Arms A and B. | 2.99 [1.66 to 4.98]
  Week 96: HOMA-IR (N=65 in C) | NA [NA to NA] — HOMA-IR was not collected at Week 96 in Arms A and B. | NA [NA to NA] — HOMA-IR was not collected at Week 96 in Arms A and B. | 2.30 [1.63 to 4.15]

15. Secondary Outcome: Sustained Virologic Response
Description: Sustained Virologic Response (SVR) was defined as undetectable HCV viral load (<60 IU/ml) 24 weeks after treatment discontinuation.
Time Frame: 24 weeks after end of treatment
Population: All Arm A, B and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Yes | 0 | 0 | 88
  No | 44 | 42 | 81

16. Secondary Outcome: Number of Participants Who Used Antianorexia Agents, Such as Megestrol and Dronabinol
Description: Use of antianorexia agents, such as megestrol and dronabinol at any time after pre-assignment.
Time Frame: Up to 96 weeks
Population: All Arm A, B and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Number of participants who used megestrol | 2 | 1 | 6
  Number of participants who used dronabinol | 4 | 4 | 22

17. Secondary Outcome: Number of Participants With Prescription as Needed of Erythropoietin (EPO), Granulocyte Colony-stimulating Factor (GCSF), and Granulocyte-monocyte Colony-stimulating Factor (GM-CSF)
Description: Prescription as needed of hematologic adjuvant therapies: erythropoietin (EPO), granulocyte colony-stimulating factor (GCSF), and granulocyte-monocyte colony-stimulating factor (GM-CSF) any time after pre-assignment
Time Frame: At any time after pre-assignment
Population: All Arm A, B and C participants
Measure: Number; unit: Participant
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
Participant
  Number of participants who used EPO | 14 | 13 | 70
  Number of participants who used GCSF | 17 | 8 | 60
  Number of participants who used GM-CSF | 0 | 0 | 0

18. Secondary Outcome: Weight
Description: Participant weight in kilograms.
Time Frame: Arms A and B: at entry and weeks 4, 8, 12, 16, 24, 32, 40, 48, 56, 64 and 72; Arm C: at entry and weeks 4, 8, 12, 16, 24, 36, 48, 72, 84 and 96.
Population: All Arm A, B and C participants who had weight available. The number of participants with results available at time points listed in the Time Frame are shown in the Data Table Row Titles below.
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | A: Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | B: OL (PEG-IFN, RBV) Then OL Randomized (Observation) | C: OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Number analyzed (Participants) | 44 | 42 | 169
kilograms
  Week 0: Weight (N=43 in A, 42 in B, 169 in C) | 74.9 [67.6 to 86.8] | 79.8 [69.7 to 88.3] | 75.8 [68.6 to 84.4]
  Week 4: Weight (N=43 in A, 35 in B, 161 in C) | 74.7 [68.6 to 87.4] | 80.4 [70.5 to 88.5] | 75.8 [68.3 to 83.5]
  Week 8: Weight (N=39 in A, 34 in B, 162 in C) | 74.9 [66.7 to 87.3] | 80.8 [71.8 to 90.9] | 75.8 [67.6 to 84.9]
  Week 12: Weight (N=42 in A, 30 in B, 157 in C) | 76.3 [67.2 to 87.9] | 81.1 [69.9 to 89.9] | 76.3 [67.4 to 83.0]
  Week 16: Weight (N=39 in A, 35 in B, 164 in C) | 77.4 [67.9 to 89.5] | 79.9 [70.0 to 90.4] | 76.3 [66.3 to 83.2]
  Week 24: Weight (N=39 in A, 36 in B, 165 in C) | 75.5 [66.3 to 89.0] | 79.4 [72.5 to 91.0] | 75.8 [65.9 to 82.6]
  Week 32: Weight (N=37 in A, 35 in B) | 76.5 [69.0 to 88.1] | 80.4 [70.8 to 87.7] | NA [NA to NA] — Weight was not collected at Week 32 in Arm C.
  Week 36: Weight (N=162 in C) | NA [NA to NA] — Weight was not collected at Week 36 in Arms A and B. | NA [NA to NA] — Weight was not collected at Week 36 in Arms A and B. | 75.0 [65.9 to 84.0]
  Week 40: Weight (N=32 in A, 29 in B) | 75.7 [67.7 to 86.4] | 83.1 [70.9 to 91.0] | NA [NA to NA] — Weight was not collected at Week 40 in Arm C.
  Week 48: Weight (N=33 in A, 31 in B, 153 in C) | 78.2 [68.8 to 88.7] | 80.4 [68.1 to 93.3] | 75.1 [66.3 to 84.4]
  Week 56: Weight (N=31 in A, 24 in B) | 79.7 [69.4 to 92.7] | 81.6 [68.8 to 90.9] | NA [NA to NA] — Weight was not collected at Week 56 in Arm C.
  Week 64: Weight (N=26 in A, 24 in B) | 78.5 [69.3 to 87.7] | 84.0 [72.8 to 91.9] | NA [NA to NA] — Weight was not collected at Week 64 in Arm C.
  Week 72: Weight (N=26 in A, 27 in B, 141 in C) | 81.6 [68.6 to 89.6] | 85.4 [71.7 to 94.0] | 75.6 [65.5 to 84.6]
  Week 84: Weight (N=140 in C) | NA [NA to NA] — Weight was not collected at Week 84 in Arms A and B. | NA [NA to NA] — Weight was not collected at Week 84 in Arms A and B. | 77.0 [67.6 to 87.6]
  Week 96: Weight (N=138) | NA [NA to NA] — Weight was not collected at Week 96 in Arms A and B. | NA [NA to NA] — Weight was not collected at Week 96 in Arms A and B. | 78.4 [69.6 to 88.0]

ADVERSE EVENTS:
Time Frame: From entry (Step 2 for Arms A and B, Step 3 for Arm C) to study completion (at Week 72 for Step 2; at week 78-84 for Step 3, depending on participants' time in Step 1).
Description: The protocol required reporting of signs/symptoms and laboratory results >=Grade 3 and events that led to a change in treatment, regardless of grade. Hemoglobin, plateles, ANC, fasting HDL, LDL and total cholesterol, insulin and glucose values were reported regardless of grade. The DAIDS AE Grading Table (1992) and Expedited AE Manual (2004) were used.
Groups:
- Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN): At week 12 (end of the initial run-in period - Step 1) participants were found to be HCV RNA positive (HCV RNA > 60 IU/mL) and had less than a 2 log decrease in HCV RNA from Baseline. For Step 2, participants were assigned to the Randomized Open Label (OL) part of the study to receive the pegylated interferon (PEG-IFN) 180 mcg weekly Arm.
- OL (PEG-IFN, RBV) Then OL Randomized (Observation): At week 12 (end of the initial run-in period - Step 1) participants were found to be HCV RNA positive (HCV RNA > 60 IU/mL) and had less than a 2 log decrease in HCV RNA from Baseline. For Step 2, participants were assigned to the Randomized Open Label (OL) part of the study to be followed on the Observation (no treatment) Arm.
- OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV): At week 12 (end of initial run-in period, Step 1) participants were found to be HCV RNA negative (HCV RNA < 60 IU/mL) or had more than a 2 log decrease in HCV RNA from Baseline. Participants were assigned to remain in the Open Label (OL) part of the study continuing the run-in treatment (PEG-IFN 180 mcg weekly & ribavirin [RBV] 1-1.2 g/day based on weight). At the beginning of week 36, participants were retested and, if found to be HCV RNA positive (HCV RNA > 60 IU/mL), participants could be randomized to OL PEG-IFN or Observation.
Arm/Group | Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) | OL (PEG-IFN, RBV) Then OL Randomized (Observation) | OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV)
Serious Adverse Events (participants affected / at risk) | 6/44 | 2/42 | 37/169
Other Adverse Events (participants affected / at risk) | 43/44 | 41/42 | 166/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) (N=44) | OL (PEG-IFN, RBV) Then OL Randomized (Observation) (N=42) | OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV) (N=169)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Death (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Neutrophil count (Investigations) | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label (OL) (PEG-IFN, RBV); OL Randomized (PEG-IFN) (N=44) | OL (PEG-IFN, RBV) Then OL Randomized (Observation) (N=42) | OL (PEG-IFN, RBV) Then OL (PEG-IFN, RBV) (N=169)
Chest pain (General disorders) | 4 | 0 | 8
Fatigue (General disorders) | 4 | 0 | 14
Pyrexia (General disorders) | 2 | 1 | 11
Bronchitis (Infections and infestations) | 2 | 0 | 9
Activated partial thromboplastin time prolonged (Investigations) | 8 | 8 | 1
Alanine aminotransferase increased (Investigations) | 30 | 32 | 64
Aspartate aminotransferase increased (Investigations) | 7 | 6 | 12
Blood bilirubin increased (Investigations) | 2 | 0 | 19
Blood glucose abnormal (Investigations) | 14 | 8 | 55
Blood glucose decreased (Investigations) | 3 | 2 | 14
Blood glucose increased (Investigations) | 11 | 7 | 16
Blood triglycerides abnormal (Investigations) | 6 | 0 | 22
Blood uric acid increased (Investigations) | 1 | 1 | 11
Gamma-glutamyltransferase increased (Investigations) | 8 | 2 | 6
Haemoglobin decreased (Investigations) | 5 | 1 | 22
Lipase increased (Investigations) | 5 | 6 | 13
Neutrophil count decreased (Investigations) | 37 | 25 | 144
Platelet count decreased (Investigations) | 21 | 9 | 58
Prothrombin time prolonged (Investigations) | 5 | 4 | 0
Weight decreased (Investigations) | 2 | 2 | 10
Depression (Psychiatric disorders) | 3 | 2 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 13
Hypertension (Vascular disorders) | 4 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve US or foreign patent or other intellectual property rights.